CLINICAL TRIAL: NCT00379301
Title: Efficacy of Different Ablation Strategies in Achieving Long-Term Arrhythmia Control in Patients With Persistent or Permanent Atrial Fibrillation
Brief Title: Efficacy of Different Ablation Strategies for Controlling Atrial Fibrillation
Acronym: RASTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPenn805173
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; A-Fib; AF; Persistent; Permanent; Pulmonary Vein Isolation; Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

ARMS (3):
- Group 1 (Active Comparator): Pulmonary vein isolation (PVI) combined with ablation of documented non-PV triggers of atrial fibrillation --- (sites away from the pulmonary veins where consistent abnormal impulses that can trigger AF are identified during the procedure)
  Interventions: Procedure: Radiofrequency ablation
- Group 2 (Active Comparator): PVI combined with ablation at documented sites of non-PV triggers, PLUS ablation at sites where non-PV triggers are commonly found
  Interventions: Procedure: Radiofrequency ablation
- Group 3 (Active Comparator): PVI combined with ablation at documented sites of non-PV triggers and ablation at sites in the left atrium that demonstrate disorganized electrical impulses called complex fractionated electrograms (CFE).
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Special catheters are inserted into blood vessels in the groin, then advanced into the left atrium of the heart. Radiofrequency (heat) energy is applied to small areas of heart tissue where electrical impulses that generate AF are found.

SUMMARY:
This study involves treatment for atrial fibrillation (AF)-the most common heart condition in the US-where the upper chambers of the heart beat very fast and in a disorganized manner. This can be felt as palpitations, tiredness, shortness of breath and passing out, plus can lead to stroke, damage to the heart muscle and a shorter life span. Study participants will receive a common treatment for atrial fibrillation called radiofrequency ablation (RFA), where small lesions or "burns" are made inside the heart to cut off the abnormal impulses that cause AF. The purpose of this study is to compare the effectiveness of three different common ablation strategies in patients with persistent or permanent AF. Subjects will be randomized (like drawing straws) to be treated with one of the three strategies to see if there is a difference in how well atrial fibrillation is controlled after treatment.

DETAILED DESCRIPTION:
In most cases, AF originates where the pulmonary veins (PV) enter the left upper chamber of the heart, known as the left atrium (LA). Common to the procedure in each arm of the study is pulmonary vein isolation (PVI) or ablation of tissue around the pulmonary vein entrances. After PVI, the procedure continues with ablation in other areas of the LA where similar abnormal impulses are found. The three strategies for continuing with ablation after PVI are described in the "Arms" section below.

ELIGIBILITY:
Inclusion Criteria:

* All patients of age ≥ 30 years, undergoing their first ablation procedure that meet ACC / AHA defined criteria for persistent or permanent AF will be eligible to participate in the study. This includes patients with a history of AF episodes lasting at least 7 days or requiring at least 2 cardioversions.

Exclusion Criteria:

1. Patients with paroxysmal AF (self-terminating episodes lasting < 7 day)
2. Patients who have had a previous AF ablation procedure
3. Pregnancy
4. Failure to obtain informed consent
5. Less than 30 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Long-term (greater than 6 months) arrhythmia control in patients with persistent or permanent AF | 6 - 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Dixit, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Dixit S, Marchlinski FE, Lin D, Callans DJ, Bala R, Riley MP, Garcia FC, Hutchinson MD, Ratcliffe SJ, Cooper JM, Verdino RJ, Patel VV, Zado ES, Cash NR, Killian T, Tomson TT, Gerstenfeld EP. Randomized ablation strategies for the treatment of persistent atrial fibrillation: RASTA study. Circ Arrhythm Electrophysiol. 2012 Apr;5(2):287-94. doi: 10.1161/CIRCEP.111.966226. Epub 2011 Dec 2. PMID 22139886